CLINICAL TRIAL: NCT00690235
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Demonstrate the Effects of Pramlintide on Weight Reduction in Clozapine- and Olanzapine-Induced Weight Gain in Obese People Diagnosed With Schizophrenia
Brief Title: Demonstrate the Effects of Pramlintide on Weight Reduction in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Carol A. Tamminga, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 092007-025
Record Dates: First submitted 2008-01-27; First posted 2008-06-04 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Diabetes; Weight Gain
Keywords: Schizophrenia; Schizoaffective; Olanzapine; Zyprexa; Clozapine; Clozaril; Pramlintide; Diabetes; Weight Gain; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Diabetes Mellitus; Weight Gain; Obesity; Metabolic Syndrome | interventions — pramlintide; Islet Amyloid Polypeptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Other): Patients will be given the Placebo for injection twice daily
  Interventions: Drug: Placebo
- Pramlintide (Other): volunteers are given 180mg of pramlintide, twice daily
  Interventions: Drug: Pramlintide

INTERVENTIONS:
Drug: Pramlintide — 180mg subcutaneous injections, twice daily
  Other Names: Amylin
  Arms: Pramlintide
Drug: Placebo — 180mg subcutaneous injections, twice daily
  Other Names: sterile saline
  Arms: Placebo

SUMMARY:
Primary Objective:

To test the effect of pramlintide on body weight in clozapine- and olanzapine-induced weight gain in persons with schizophrenia who are currently taking either drug; measures of the metabolic syndrome will be evaluated as well.

DETAILED DESCRIPTION:
This study is a sixteen week placebo-controlled, double-blind investigation of the effect of pramlintide on body weight in clozapine- and olanzapine-induced weight gain. We will recruit approximately 72 volunteers with the plan of having a final N = 25 in each of the 2 treatment groups. (This number is to allow for normal attrition in this patient population. If needed, we will recruit more than 72 volunteers in order to achieve the appropriate number of completed subjects.) Patients will be recruited from the local Dallas public and VA mental health systems as volunteers for this study. This study is anticipated to last 20 weeks (2 weeks lead-in [approximately 2-3 visits], 1 week training [4 visits], 16 weeks active drug/placebo [one visit per week for the first 4 weeks, then one visit every 2 weeks for the remainder], and one week follow-up [one visit]. Please see attached chart for more details about each visit.) Volunteers will have to have a history of significant weight gain accompanying olanzapine or clozapine treatment and have a BMI=>27 and =<40. Each volunteer will be maintained on their optimal dose of clozapine or olanzapine and be randomized blindly to pramlintide or placebo. Pramlintide will be administered by the patients in a self-injectable form and dosing will begin at 180 mcg bid for 2 weeks and then increase to 360 mcg bid for the remainder of the study. The randomization to pramlintide/placebo will be preceded by a week-long self-administration training program using placebo for pramlintide (with additional information regarding nutrition, exercise, general self-care, and risk factors for diabetes being provided to the patients during this training program).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers will be males or females 18-65 yrs of age with a diagnosis of schizophrenia or schizoaffective disorder who have a history of significant weight gain with olanzapine or clozapine administration.
* Volunteers will have a current BMI=>27 but equal to or less than 40.
* Volunteers will have been taking a stable dose (less than 10% dose change) of clozapine or olanzapine or at least two months prior to study start.
* Volunteers will be willing and able to participate in the subcutaneous administration training week prior to study start.
* Able and willing to give informed consent.

Exclusion Criteria:

* Clinically significant abnormal pre-admission vital signs, positive HIV, or clinical laboratory evaluations, in which the principal investigator deems the subject-volunteer ineligible for the study

  * Positive results for infectious diseases and sexually-transmitted diseases will be reported according to the Texas Department of State Health and Texas Administrative Code rules and guidelines
* Any patient with current diabetes mellitus, even if caused by antipsychotic use .
* Patients with active liver disease requiring current treatment. Positive hepatitis C volunteers will only be excluded if they have active liver disease or they have enzyme values are two times the upper limit of normal.
* Any patients with medical disorders that are not properly controlled by medications.
* Pregnant women or women who are breast feeding.
* Patients concomitantly treated with another conventional or second generation antipsychotic medication or with any other anti-obesity drug.
* Mental capacity is limited to the extent that the patient cannot understand the nature of the study along with its risks and benefits.
* Subjects with a high risk of suicide since there is a potential that the study medication will lower the subject's glucose levels.
* Any patient judged by the principal investigator to be inappropriate for the study.
* Known hypersensitivity to study medication or its components
* Non-English speaking

  * The clinical assessments that will be used are not available in valid and reliable forms for non-English speaking populations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Tamminga, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients will be given the Placebo for injection twice daily
  Placebo: 180mg subcutaneous saline injections, twice daily
Period: Overall Study
Arm/Group | Pramlintide | Placebo
Started | 17 | 16
Completed | 12 | 12
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramlintide | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss With Pramlintide in Persons With Schizophrenia Who Have Gained Weight Taking Olanzapine or Clozapine
Description: Mean Number of Pounds Lost on Pramlintide Over 16 Weeks
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- Placebo: Volunteers will be given the Placebo for injection twice daily
  Placebo: 180mg subcutaneous injections, twice daily
Arm/Group | Pramlintide | Placebo
Number analyzed (Participants) | 12 | 12
pounds | 37 (143.06) | 40.5 (109.26)

ADVERSE EVENTS:
Arm/Group | Pramlintide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pramlintide (N=12) | Placebo (N=12)
Pain/bruise at injection site (Psychiatric disorders) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No